CLINICAL TRIAL: NCT03446781
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Of EN3835 In The Treatment Of Edematous Fibrosclerotic Panniculopathy (Cellulite)
Brief Title: Effectiveness and Safety of EN3835 in the Treatment of Cellulite in Women
Acronym: RELEASE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EN3835-303
Record Dates: First submitted 2018-02-04; First posted 2018-02-27 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Edematous Fibrosclerotic Panniculopathy (Cellulite)
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EN3835 Active (Active Comparator): EN3835 0.84mg (Collagenase Clostridium Histolyticum)
  Interventions: Biological: EN3835
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: EN3835 — Collagenase clostridium histolyticum
  Arms: EN3835 Active
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Subjects will be screened for study eligibility within 14 days prior to enrolling in this study. Subjects with 2 treatment areas (bilateral buttocks) with moderate or severe levels of cellulite as independently assessed by the subject using the Patient Reported Photonumeric Cellulite Severity Scale (PR-PCSS) and by the Investigator using the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS) will be eligible. The eligibility of the buttocks will be confirmed on Day 1. Once the eligibility of the buttocks is confirmed, subjects will be randomly assigned to a treatment group (EN3835 0.84 mg per buttock or placebo) in a 1:1 ratio within an investigational site. Each subject will receive a treatment course which consists of up to 3 treatment visits (sessions), separated by 21 days (ie, Days 1, 22, and 43). Each treatment visit will consist of 12 injections (0.3 mL per injection of EN3835 0.07 mg/injection or placebo; 0.84 mg in 3.6 mL per buttock) in each of the two buttocks for a total volume of 7.2 mL (1.68 mg). Selection of dimples to be treated in the buttocks will be at the discretion of the Investigator. End of study will occur at study day 71.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date an informed consent agreement
2. Be a female ≥18 years of age
3. At Screening visit, have 2 bilateral buttocks with each buttock having:

   1. a score of 3 or 4 (moderate or severe) as reported by the subject (PR-PCSS), and
   2. a score of 3 or 4 (moderate or severe) as reported by the Investigator (CR-PCSS)
4. At Day 1 visit, have 2 bilateral buttocks with each buttock having:

   1. a score of 3 or 4 (moderate or severe) as reported by the subject (PR-PCSS), and
   2. a score of 3 or 4 (moderate or severe) as reported by the Investigator (CR-PCSS)
5. Be willing to apply sunscreen to the buttocks before each exposure to the sun while participating in the study (ie, Screening through end of study)
6. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at Screening
7. Have a negative serum pregnancy test at Screening and a negative urine pregnancy test before injection of study drug and be using a stable and effective contraception method (eg, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or double barrier method) for at least 1 menstrual cycle prior to study enrollment and for the duration of the study; or be menopausal defined as 12 months of amenorrhea in the absence of other biological or physiological causes, as determined by the Investigator; or post-menopausal for at least 1 year; or be surgically sterile
8. Be willing and able to cooperate with the requirements of the study
9. Be able to read, complete and understand the patient-reported outcomes rating instruments in English

Exclusion Criteria:

1. Has any of the following systemic conditions:

   1. Coagulation disorder
   2. Evidence or history of malignancy (other than excised basal-cell carcinoma) unless there has been no recurrence in at least 5 years
   3. History of keloidal scarring or abnormal wound healing
   4. Concurrent diseases or conditions that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. Any questions about concurrent diseases should be discussed with the Medical Monitor
   5. Evidence of clinically significant abnormalities on physical examination, vital signs, electrocardiogram (ECG), or clinical laboratory values
2. Has any of the following local conditions in the areas to be treated:

   1. History of lower extremity thrombosis or post-thrombosis syndrome
   2. Vascular disorder (eg, varicose veins, telangiectasia) in area to be treated
   3. Inflammation or active infection
   4. Severe skin laxity, flaccidity, and/or sagging
   5. Active cutaneous alteration including rash, eczema, psoriasis, or skin cancer
   6. Has a tattoo and/or a mole located within 2 cm of the site of injection
3. Requires the following concomitant medications before or during participation in the trial:

   a. Anticoagulant or antiplatelet medication or has received anticoagulant or antiplatelet medication (except for ≤150 mg aspirin daily) within 7 days before injection of study drug
4. Has used any of the following for the treatment of EFP on a buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:

   1. Liposuction in a buttock during the 12-month period before injection of study drug
   2. Injections (eg, mesotherapy); radiofrequency device treatments; laser treatment; buttock implant treatment; cryolipolysis; or surgery (including subcision and/or powered subcision) within a buttock during the 12-month period before injection of study drug
   3. Any investigational treatment for EFP on a buttock during the 12-month period before the injection of study drug
   4. Endermologie or similar treatments within a buttock during the 6-month period before injection of study drug
   5. Massage therapy within a buttock during the 3-month period before injection of study drug
   6. Creams (eg, Celluvera™, TriLastin®) and/or home therapies to prevent or mitigate EFP within a buttock during the 2-week period before injection of study drug
5. Is presently nursing or providing breast milk
6. Intends to become pregnant during the study
7. Intends to initiate an intensive sport or exercise program during the study
8. Intends to initiate a weight reduction program during the study
9. Intends to use tanning spray or tanning booths during the study
10. Has received an investigational drug or treatment within 30 days before injection of study drug
11. Has a known systemic allergy to collagenase or any other excipient of study drug
12. Has received any collagenase treatments at any time prior to treatment
13. Was a subject in a previous cellulite clinical trial of CCH: AUX-CC-830, AUX-CC-831, EN3835-102, EN3835-104, EN3835-201, EN3835-202, and/or EN3835-205
14. Any other condition(s) that, in the Investigator's opinion, might indicate the subject to be unsuitable for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McLane, Study Director — Endo Pharmaceuticals
Locations (25):
- United States (25):
  - Endo Clinical Trial Site #1, Glendale, Arizona
  - Endo Clinical Trial Site #2, North Little Rock, Arkansas
  - Endo Clinical Trial Site #3, Beverly Hills, California
  - Endo Clinical Trial Site #4, Murrieta, California
  - Endo Clinical Trial Site #5, Newport Beach, California
  - Endo Clinical Trial Site #6, San Diego, California
  - Endo Clinical Trial Site #7, Greenwood Village, Colorado
  - Endo Clinical Trial Site #8, Coral Gables, Florida
  - Endo Clinical Trial Site #9, Miami, Florida
  - Endo Clinical Trial Site #10, Nampa, Idaho
  - Endo Clinical Trial Site #11, Carmel, Indiana
  - Endo Clinical Trial Site #12, Metairie, Louisiana
  - Endo Clinical Trial Site #13, New Orleans, Louisiana
  - Endo Clinical Trial Site #14, Warren, Michigan
  - Endo Clinical Trial Site #15, Montclair, New Jersey
  - Endo Clinical Trial Site #16, East Setauket, New York
  - Endo Clinical Trial Site #17, New York, New York
  - Endo Clinical Trial Site #18, Cincinnati, Ohio
  - Endo Clinical Trial Site #19, Nashville, Tennessee
  - Endo Clinical Trial Site #20, Austin, Texas
  - Endo Clinical Trial Site #21, Beaumont, Texas
  - Endo Clinical Trial Site #22, Houston, Texas
  - Endo Clinical Trial Site #23, San Antonio, Texas
  - Endo Clinical Trial Site #24, Salt Lake City, Utah
  - Endo Clinical Trial Site #25, Lynchburg, Virginia

REFERENCES:
- [Derived] Kaufman-Janette J, Joseph JH, Kaminer MS, Clark J, Fabi SG, Gold MH, Goldman MP, Katz BE, Peddy K, Schlessinger J, Young VL, Davis M, Hurley D, Liu G, McLane MP, Vijayan S, Bass LS. Collagenase Clostridium Histolyticum-aaes for the Treatment of Cellulite in Women: Results From Two Phase 3 Randomized, Placebo-Controlled Trials. Dermatol Surg. 2021 May 1;47(5):649-656. doi: 10.1097/DSS.0000000000002952. PMID 33840781

RESULTS

PARTICIPANT FLOW:
Groups:
- Collagenase Clostridium Histolyticum (CCH): CCH 0.84 mg/Buttock 1.68 mg Total Dose
- Placebo: Placebo-control
Period: Overall Study
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Started | 214 | 208
Completed | 186 | 191
Not Completed | 28 | 17
Not completed — Lost to Follow-up | 11 | 5
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Adverse Event | 8 | 2
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo | Total
Number analyzed (Participants) | 214 | 206 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.62) | 45.7 (11.16) | 46.7 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 206 | 420
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 58 | 104
  Not Hispanic or Latino | 168 | 148 | 316
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 32 | 61
  White | 179 | 164 | 343
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 2 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.52 (6.184) | 31.14 (7.567) | 30.82 (6.896)
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale White) | 6 | 8 | 14
  II (Fair) | 74 | 54 | 128
  III (Darker White) | 50 | 64 | 114
  IV (Light Brown) | 53 | 47 | 100
  V (Brown) | 15 | 18 | 33
  VI (Dark Brown) | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: 2-level Composite Responders for the Target Buttock
Description: Proportion of 2-level Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) / Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) composite responders in the target buttock at Day 71. CR-PCSS and PR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe). A 2-level composite responder is defined as a participant with improvement from baseline of at least 2-levels of severity in the CR-PCSS and an improvement from baseline of at least 2-levels of severity in the PR-PCSS of the target buttock. A participant who missed one or two assessments of CR-PCSS and PR-PCSS at Day 71 was defined as a non-responder.
Time Frame: Day 71
Population: ITT Population includes all randomized participants who had at least 1 injection of study drug. All demographic and baseline characteristic summaries were based on this population. The primary and key secondary efficacy parameters were summarized based on this population.
Measure: Count of Participants; unit: Participants
Groups:
- Collagenase Clostridium Histolyticum (CCH): CCH 0.84 mg/Buttock
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants
  Yes | 12 | 1
  No | 202 | 205
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Adjusted for analysis center

2. Secondary Outcome: 1-level PR-PCSS Responders of the Target Buttock
Description: Improvement in cellulite severity of the Target Buttock from baseline of at least 1-level of severity in Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS). PR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe).
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants
  Yes | 124 | 61
  No | 90 | 145
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

3. Secondary Outcome: 2-level PR-PCSS Responders of the Target Buttock
Description: Improvement in cellulite severity of the Target Buttock from baseline of at least 2-levels of severity in Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS). PR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe).
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants
  Yes | 45 | 12
  No | 169 | 194
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

4. Secondary Outcome: 1-level Composite Responders of the Target Buttock
Description: Improvement in cellulite severity of the Target Buttock from baseline of at least 1-level of severity in Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) / Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS). PR-PCSS and CR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe).
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants
  Yes | 89 | 23
  No | 125 | 183
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

5. Secondary Outcome: 2-level Composite Responders of the Non-target Buttock
Description: Improvement in cellulite severity of the Non-target Buttock from baseline of at least 2-levels of severity in Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) / Clinician -Reported Photonumeric Cellulite Severity Scale (CR-PCSS). PR-PCSS and CR-PCSS is a 5-level scale ranging from "0" (None) to "4" (Severe).
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants
  Yes | 13 | 4
  No | 201 | 202
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p = 0.033, Cochran-Mantel-Haenszel; Adjusted for analysis center

6. Secondary Outcome: 1-level SSRS Responders
Description: Subject Self-Rating Scale (SSRS) is a measure that assesses participant satisfaction with appearance in association with cellulite on the buttocks using whole numbers on a 7-level scale that ranges from "0" (Extremely Dissatisfied) to "6" (Extremely Satisfied). A 1-level SSRS responder is defined as a participant who is at least slightly satisfied (Slightly Satisfied [4], Very Satisfied [5], or Extremely Satisfied [6]) with the appearance of the cellulite on her buttocks at Day 71.
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Collagenase Clostridium Histolyticum (CCH): CCH 0.84 mg/Buttock (1.68 mg Total Dose)
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants | 90 | 31
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

7. Secondary Outcome: Change From Baseline in PR-CIS Total Score
Description: Patient-Reported Cellulite Impact Scale (PR-CIS) is a 6-item static questionnaire, each item is answered by a participant on a 11-level numerical rating scale that ranges from "0" (Not at all) to "10" (Extremely). The PR-CIS total score is the sum of individual item scores and can range from "0" to "60" with higher numbers reflecting a more negative impact from the cellulite. A responder is defined as a participant with a reduction in the PR-CIS total score of at least 12 from baseline at evaluation time point. A negative change from baseline indicates an improvement in cellulite severity.
Time Frame: Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
score on a scale
  Baseline (Day 1): number analyzed (Participants) | 213 | 202
  Baseline (Day 1) | 52.4 (8.01) | 51.6 (9.40)
  Day 71 | 40.9 (13.57) | 45.1 (12.65)
  Change from Baseline: number analyzed (Participants) | 213 | 202
  Change from Baseline | -11.5 (12.74) | -6.5 (11.74)
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, ANCOVA; With factors of treatment group and analysis center adjusted for baseline values in the model

8. Secondary Outcome: 1-level S-GAIS Responders of Target Buttock
Description: Subject Global Aesthetic Improvement Scale (S-GAIS) is a measure that assesses participant rating of cellulite appearance after treatment. This scale has 7-levels ranging from "+3" (Very Much Improved) to "-3" (Very Much Worse). Responders are defined as participants with ≥1-level improvement (Improved, Much Improved or Very Improved) in S-GAIS assessment of the Target Buttock.
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants | 126 | 46
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

9. Secondary Outcome: 2-level S-GAIS Responders of Target Buttock
Description: Subject Global Aesthetic Improvement Scale (S-GAIS) is a measure that assesses participant rating of cellulite appearance after treatment. This scale has 7-levels ranging from "+3" (Very Much Improved) to "-3" (Very Much Worse). Responders are defined as participants with ≥ 2-level improvement (Much Improved or Very Much Improved) in S-GAIS assessment of the Target Buttock.
Time Frame: Day 71
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
Number analyzed (Participants) | 214 | 206
Participants | 38 | 9
Statistical Analysis 1: Comparison: Collagenase Clostridium Histolyticum (CCH) vs Placebo; CCH 0.84 mg/Buttock versus Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for analysis center

10. Secondary Outcome: PR-PCSS Rating for the Target and Non-target Buttock by Visit
Description: The Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level photonumeric scale used by the patient (participant) to assess the severity of the participant's cellulite. The ratings range from "0" (None) to "4" (Severe).
Time Frame: Day 71
Population: mITT Population includes all ITT participants with a baseline and at least 1 post-injection evaluation of both the CR-PCSS and PR-PCSS for both the target and non-target buttocks. All secondary and supportive efficacy evaluations were based on the mITT Population.
Measure: Count of Participants; unit: Participants
Groups:
- Day 1: CCH: Baseline (Day 1) for CCH Treated Group
- Day 1: Placebo: Baseline (Day 1) for PlaceboGroup
- Day 22: CCH: Day 22 for CCH Treated Group
- Day 22: Placebo: Day 22 for Placebo Group
- Day 43: CCH: Day 43 for CCH Treated Group
- Day 43: Placebo: Day 43 for Placebo Group
- Day 71: CCH: Day 71 for CCH Treated Group
- Day 71: Placebo: Day 71 for Placebo Group
- Day 71: CCH (LOCF): Day 71 for CCH Treated Group (Last Observation Carried Forward)
- Day 71: Placebo (LOCF): Day 71 for Placebo Group (Last Observation Carried Forward)
Arm/Group | Day 1: CCH | Day 1: Placebo | Day 22: CCH | Day 22: Placebo | Day 43: CCH | Day 43: Placebo | Day 71: CCH | Day 71: Placebo | Day 71: CCH (LOCF) | Day 71: Placebo (LOCF)
Number analyzed (Participants) | 209 | 201 | 209 | 201 | 209 | 201 | 209 | 201 | 209 | 201
Participants
  Target Buttock Rating: number analyzed (Participants) | 209 | 201 | 197 | 199 | 186 | 191 | 186 | 191 | 209 | 201
  Target Buttock Rating: None (0) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0
  Target Buttock Rating: Almost None (1) | 0 | 0 | 1 | 1 | 17 | 3 | 19 | 2 | 19 | 2
  Target Buttock Rating: Mild (2) | 0 | 0 | 45 | 17 | 61 | 26 | 61 | 32 | 64 | 32
  Target Buttock Rating: Moderate (3) | 89 | 82 | 78 | 79 | 67 | 85 | 65 | 76 | 76 | 81
  Target Buttock Rating: Severe (4) | 120 | 119 | 73 | 101 | 41 | 77 | 38 | 81 | 47 | 86
  Non-target Buttock Rating: number analyzed (Participants) | 209 | 201 | 197 | 199 | 186 | 191 | 186 | 191 | 209 | 201
  Non-target Buttock Rating: None (0) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Non-target Buttock Rating: Almost None (1) | 0 | 0 | 3 | 0 | 17 | 4 | 21 | 3 | 21 | 3
  Non-target Buttock Rating: Mild (2) | 0 | 0 | 38 | 19 | 55 | 24 | 58 | 32 | 64 | 34
  Non-target Buttock Rating: Moderate (3) | 96 | 71 | 82 | 71 | 67 | 86 | 66 | 72 | 74 | 75
  Non-target Buttock Rating: Severe (4) | 113 | 130 | 74 | 108 | 47 | 77 | 40 | 84 | 49 | 89

11. Secondary Outcome: Subjects Satisfaction With Cellulite Treatment
Description: A 1-level Subject Satisfaction Responder is defined as a participant who is at least satisfied (Satisfied [+1], or Very Satisfied [+2]) with the appearance of the cellulite on her buttocks at the Day 71 visit. A positive change indicates an improvement in cellulite.
Time Frame: Day 71
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Day 71: CCH | Day 71: Placebo | Day 71: CCH (LOCF) | Day 71: Placebo (LOCF)
Number analyzed (Participants) | 186 | 191 | 198 | 195
Participants
  Very Satisfied (+2) | 15 | 4 | 15 | 4
  Satisfied (+1) | 72 | 22 | 74 | 22
  Neither Satisfied Nor Dissatisfied (0) | 60 | 73 | 64 | 75
  Dissatisfied (-1) | 24 | 47 | 29 | 48
  Very Dissatisfied (-2) | 15 | 45 | 16 | 46

12. Other Pre Specified Outcome: Serum Antibody Positivity by Visit
Description: Percent of participants that are seropositive. Percentages were based on the number of subjects who had immunogenicity lab samples analyzed at the visit.
Time Frame: Day 1 - Day 71
Population: Safety Population includes all participants who received at least 1 dose of CCH in this study. All safety parameters were summarized based on this population.
Measure: Count of Participants; unit: Participants
Groups:
- Anti-AUX-I: CCH: Antibody AUX-I for the CCH Treated Group
- Anti-AUX-I: Placebo: Antibody AUX-I for the Placebo Group
- Anti-AUX-II: CCH: Antibody AUX-II for the CCH Treated Group
- Anti-AUX-II: Placebo: Antibody AUX-II for the Placebo Group
Arm/Group | Anti-AUX-I: CCH | Anti-AUX-I: Placebo | Anti-AUX-II: CCH | Anti-AUX-II: Placebo
Number analyzed (Participants) | 214 | 206 | 214 | 206
Participants
  Day 1: Seropositive | 6 | 2 | 3 | 6
  Day 1: Seronegative | 208 | 204 | 211 | 200
  Day 22: number analyzed (Participants) | 196 | 199 | 196 | 199
  Day 22: Seropositive | 106 | 1 | 52 | 7
  Day 22: Seronegative | 90 | 198 | 144 | 192
  Day 43: number analyzed (Participants) | 186 | 190 | 186 | 190
  Day 43: Seropositive | 183 | 4 | 183 | 7
  Day 43: Seronegative | 3 | 186 | 3 | 183
  Day 71: number analyzed (Participants) | 186 | 190 | 186 | 190
  Day 71: Seropositive | 186 | 8 | 185 | 9
  Day 71: Seronegative | 0 | 182 | 1 | 181

13. Other Pre Specified Outcome: Overall Antibody Titer Levels by Visit
Description: Descriptive statistics were based on log10 transformation of titer levels. Titer levels were imputed as 10 before the transformation if the reported level is "<10". Only seropositive participants are summarized.
Time Frame: Day 1 - Day 71
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: log 10 titer
Arm/Group | Anti-AUX-I: CCH | Anti-AUX-I: Placebo | Anti-AUX-II: CCH | Anti-AUX-II: Placebo
Number analyzed (Participants) | 214 | 206 | 214 | 206
log 10 titer
  Day 1 positive: number analyzed (Participants) | 6 | 2 | 3 | 6
  Day 1 positive | 2.235 (1.7365) | 1.000 (0.0000) | 3.212 (0.8056) | 1.365 (0.3834)
  Day 22 positive: number analyzed (Participants) | 106 | 1 | 52 | 7
  Day 22 positive | 2.331 (1.2566) | 3.504 | 1.912 (1.2718) | 1.387 (0.4788)
  Day 43 positive: number analyzed (Participants) | 183 | 4 | 183 | 7
  Day 43 positive | 4.602 (0.8721) | 2.539 (1.1462) | 3.680 (1.0617) | 1.302 (0.4596)
  Day 71 positive: number analyzed (Participants) | 186 | 8 | 185 | 9
  Day 71 positive | 5.898 (0.7131) | 2.039 (1.2854) | 5.255 (0.7142) | 1.572 (0.7895)

14. Other Pre Specified Outcome: Presence of Neutralizing Antibody (Seropositivity) at Day 71 (LOCF) by Antidrug Antibody Log Titer Quartiles
Description: Q1 and Q4 are based on the ADA titer levels.
Time Frame: Day 71
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- CCH: Q1: Q1 for the CCH Treated Group
- CCH: Q4: Q4 for the CCH Treated Group
- CCH: Total: Total CCH
Arm/Group | CCH: Q1 | CCH: Q4 | CCH: Total
Number analyzed (Participants) | 24 | 24 | 48
Participants
  Neutralizing AUX-I Antibody: Negative | 12 | 3 | 15
  Neutralizing AUX-I Antibody: Positive | 12 | 21 | 33
  Neutralizing AUX-II Antibody: Negative | 5 | 1 | 6
  Neutralizing AUX-II Antibody: Positive | 19 | 23 | 42

ADVERSE EVENTS:
Time Frame: All (serious and nonserious) AEs, from Day 1 to Day 71
Description: All (serious and nonserious) AEs, whether elicited or observed during study visits or spontaneously reported by the participant, including events that occurred from the time the participant signed the study-specific consent form until completion of or discharge from the study.
Arm/Group | Collagenase Clostridium Histolyticum (CCH) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/206
Serious Adverse Events (participants affected / at risk) | 1/214 | 0/206
Other Adverse Events (participants affected / at risk) | 203/214 | 64/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Collagenase Clostridium Histolyticum (CCH) (N=214) | Placebo (N=206)
Syncope (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Collagenase Clostridium Histolyticum (CCH) (N=214) | Placebo (N=206)
Injection site bruising (General disorders) | 193 | 42
Injection site pain (General disorders) | 127 | 26
Injection site nodule (General disorders) | 70 | 2
Injection site pruritus (General disorders) | 34 | 3
Injection site erythema (General disorders) | 28 | 17
Injection site discolouration (General disorders) | 21 | 2
Injection site mass (General disorders) | 15 | 0
Injection site warmth (General disorders) | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03446781/Prot_SAP_000.pdf